CLINICAL TRIAL: NCT05100017
Title: Methocarbamol vs Oxybutynin for Management of Pain and Discomfort S/P Ureteroscopy Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Professor of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00214901
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Kidney Calculi; Kidney Diseases; Nephrolithiasis; Urolithiasis; Ureteral Diseases; Ureteral Calculi
MeSH Terms: conditions — Kidney Calculi; Kidney Diseases; Nephrolithiasis; Urolithiasis; Ureteral Diseases; Ureteral Calculi | interventions — Methocarbamol; oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methocarbamol (Active Comparator): Patients will receive oral Methocarbamol 750mg every six hours after ureteroscopy as needed for pain in addition to the standard postoperative pain regimen (Tylenol 1000mg every six hours, Tamsulosin 0.4mg daily, phenazopyridine 200mg every eight hours, and diclofenac 50mg every eight hours).
  Interventions: Drug: Methocarbamol
- Oxybutynin (Active Comparator): Patients will receive oral Oxybutynin XL 10mg daily after ureteroscopy as needed for pain in addition to the standard postoperative pain regimen (Tylenol 1000mg every six hours, Tamsulosin 0.4mg daily, phenazopyridine 200mg every eight hours, and diclofenac 50mg every eight hours).
  Interventions: Drug: Oxybutynin

INTERVENTIONS:
Drug: Methocarbamol — Patients will receive oral Methocarbamol 750mg every six hours as needed for pain post ureteroscopy in addition to the standard postoperative pain regimen.
  Arms: Methocarbamol
Drug: Oxybutynin — Patients will receive oral Oxybutynin XL 10mg daily for pain post ureteroscopy in addition to the standard postoperative pain regimen.
  Arms: Oxybutynin

SUMMARY:
Stone disease is a common condition, affecting approximately 9% of Americans in 2007. It causes great morbidity and is also a costly condition, estimated to cost the US healthcare system approximately 3.79 billion dollars in 2007. Ureteroscopy (URS) is the most commonly performed surgical treatment for upper tract stone disease. Ureteral stenting is a common practice after ureteroscopy and placed in ~75% of cases to prevent ureteral edema and renal obstruction. Unfortunately, ureteral stenting can be very painful and has been shown to increase the rate of emergency room visits. Many strategies have been attempted to decrease pain with ureteral stenting including modification of stent material and designs, but efforts so far have been unsuccessful in decreasing stent-related morbidity. Stent-related morbidity is hypothesized to be secondary to irritation of ureteral/bladder mucosa and muscle. Analgesics such as alpha blockers and NSAIDs have been shown to reduce stent morbidity. Anticholinergic drugs are also utilized as they decrease bladder spasms and, therefore, are hypothesized to reduce stent irritation. However, the evidence for anticholinergics has been conflicting. Anticholinergics also have a serious side effect profile including dry mouth, dry eyes, constipation, urinary retention, blurred vision, and even dementia. Some authors even hypothesize that these side effects may offset any purported benefits the anticholinergics provide for stent-morbidity.

Methocarbamol is anti-spasmodic muscle relaxant that is believed to work by acting on central neurons and possibly by blocking sodium channels. Given that anticholinergics have many side effects and questionable efficacy, the investigators hypothesize that methocarbamol may achieve superior analgesia for stent morbidity and stent-related bladder spasms.

Oxybutynin is used for the treatment of overactive bladder. The rationale is that the oxybutynin relaxes the muscles in the bladder to help decrease problems of urgency and frequent urination caused by the urinary stent irritation. Since anticholinergics have multiple side effects, finding an equally efficacious alternative with less side effects is highly desirable.

This study will evaluate the clinical and demographic factors of patients undergoing ureteroscopy and treated postoperatively with methocarbamol vs. oxybutynin for stent-related morbidity. Additionally, the study will aim to understand the postoperative outcomes and complication rates of patients discharged with methocarbamol vs. oxybutynin after ureteroscopy with a ureteral stent in place.

DETAILED DESCRIPTION:
This study is comparing the effectiveness of pain control after ureteroscopy for stone removal between two medications: oral Oxybutynin XL 10mg daily and oral Methocarbamol 750mg every six hours as needed for spasms. The study medications will be given in addition to a standard postoperative pain regiment including Tylenol 1000mg every six hours, Tamsulosin 0.4mg daily, phenazopyridine 200mg every eight hours, and diclofenac 50mg every eight hours, and finally the investigational agent (either oral oxybutynin XL 10mg once daily or oral methocarbamol 750mg every six hours as needed for pain depending on which group the participant is randomly assigned).

Patients who will be undergoing ureteroscopy for stone removal (anyone with upper tract stones, total stone burden < 2 cm) will be identified in clinic and consented to participate in the study. Patients will be randomized to either methocarbamol or oxybutynin in a 1:1 fashion using RedCAP prior to the procedure. Pain regimen after surgery includes: Tylenol 1000mg every six hours, Tamsulosin 0.4 mg daily, phenazopyridine 200mg every eight hours, and diclofenac 50mg every eight hours, and finally the investigational agent (either oral oxybutynin XL 10 mg once daily or oral methocarbamol 750mg every six hours as needed for pain). Both drugs are FDA approved, but will be used off-label for the purposes of this study. Although oxybutynin is not FDA approved for the treatment of ureteral spasms, multiple studies have been performed to study its efficacy for this indication and it will be used in an off-label fashion. The study will document age, sex, BMI, preoperative stone burden, laterality of surgery, OR duration, laser energy (kJ), laser settings, ureteral access sheath use, stent size, stent duration, stone analysis, preoperative urine culture, stone culture, and any medical comorbidities. Neither patients nor investigators will be blinded to which drug they are receiving.

Patients will be administered the PROMIS questionnaire, which has been validated for assessing ureteral stent symptoms. The VAS pain scale will also be administered to assess pain (scores from 1-10). The PROMIS questionnaire and VAS pain scale will be administered at time of study enrollment or prior to surgery. The questionnaire and VAS pain scale will be administered daily by text message (RedCAP electronic survey) from POD1 until the day of stent removal, and 1 day after the stent is removed. Stent removal typically occurs 3-7 days after surgery. The questionnaires will be completed by the patient on a mobile device. Patients will be asked to complete a drug diary, so study investigators can ensure they took the medication as prescribed. On the final survey (the one sent 1day after stent removal), the study investigators will also inquire about if the patient had any unplanned clinic or ED visits during the period the stent was in.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between age 18-80 years who are diagnosed with stones who undergo ureteroscopy and ureteral stent placement.
2. Patients who consent to the procedure will be randomized in 1:1 fashion by RedCAP either to the methocarbamol or oxybutynin arm. All patients will receive standard of care diclofenac, tamsulosin, and pyridium for pain control plus one of the study drugs.
3. Willing to take only diclofenac (or tramadol for patients with contraindication to diclofenac), phenazopyridine, and acetaminophen for post stent placement discomfort.
4. Willing to sign the Informed Consent Form.
5. Able to read, understand, and complete patient questionnaires, pain texts, and medication diary.

Exclusion Criteria:

1. Active, symptomatic urinary tract infection.
2. Non-stone related ureteral obstruction or stricture.
3. Procedural trauma or significant retained stone burden that could significantly contribute to patient discomfort.
4. Spinal cord injuries (sensory loss due to injury).
5. Non-stone related voiding dysfunction requiring supplemental bladder drainage tubes for more than 24 hours post operatively.
6. Chronic opioid usage for pain.
7. Members of vulnerable patient populations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient discomfort/pain after ureteroscopy and ureteral stent placement | 1 week
  Patients will be administered the VAS pain scale to assess pain scores (score from 1-10). The VAS pain scale will be administered at the time of study enrollment, daily from POD1 until the day of stent removal, and 1 day after the stent is removed.
Patient ureteral stent symptoms after ureteroscopy and ureteral stent placement | 1 week
  Patients will be administered the PROMIS questionnaire, which has been validated for assessing ureteral stent symptoms. The questionnaire will be administered at the time of study enrollment, daily from POD1 until the day of stent removal, and 1 day after the stent is removed.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States